CLINICAL TRIAL: NCT01437267
Title: A Phase 2, Randomized, Controlled, Observer Blind, Single Center Study of the Safety, Reactogenicity and Immunogenicity of the NVGH Glycoconjugate Vaccine Against S. Typhi in Children, Older Infants and Infants
Brief Title: Safety and Immunogenicity of Vi-CRM197 Vaccine Against S. Typhi in Children, Older Infants and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H01_05TP
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Results first posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-03

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine; Polysaccharides; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Vi-CRM, Older infants (Experimental): Older Infants (9 to 12 months) receiving 2 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- PNC13, Older infants (Active Comparator): Older infants (9 to 12 months) receiving 2 doses of Pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine
- Vi-CRM, Infants (Experimental): Infants (6 to 8 weeks) receiving 3 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- PNC13, Infants (Active Comparator): Infants (6 to 8 weeks) receiving 3 doses of Pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine
- Vi-CRM, Children (Experimental): Children (24 to 59 months) receiving 2 doses of NVGH Vi-CRM197 vaccine
  Interventions: Biological: Vi-CRM197 vaccine
- Vi-PS, Children (Active Comparator): Children (24 to 59 months) receiving 1 dose of licensed Vi Polysaccharide vaccine and 1 dose of Pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine; Biological: Vi Polysaccharide (PS) vaccine

INTERVENTIONS:
Biological: Vi-CRM197 vaccine
  Arms: Vi-CRM, Children; Vi-CRM, Infants; Vi-CRM, Older infants
Biological: Pneumococcal conjugate vaccine
  Other Names: Prevenar 13
  Arms: PNC13, Infants; PNC13, Older infants; Vi-PS, Children
Biological: Vi Polysaccharide (PS) vaccine
  Other Names: Typherix
  Arms: Vi-PS, Children

SUMMARY:
This phase 2 trial is aimed to obtain information on the safety and immunogenicity of the Vi-CRM197 in children and infants from various age groups in the Philippines where Typhoid Fever is highly endemic and an efficacious vaccine against this disease is very much needed.

ELIGIBILITY:
Inclusion criteria:

* Subjects belonging to 3 age groups will be enrolled into the trial: children (24 to 59 months of age at enrollment), older infants (9 to 12 months of age at enrollment) and infants (6 weeks of age at enrolment).
* Written informed consent will be obtained by the parents/ guardians before enrollment into the trial.
* Infants who have been vaccinated with BCG and HBV at birth and OPV at any time since birth can be enrolled into the trial, while infants who have received DTwP+HBV+Hib due at 6 weeks of age as per local EPI schedule cannot be enrolled into the trial.

Ages: 6 Weeks to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2011-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rosario Z Capeding, MD, Principal Investigator — Research Institute for Tropical Medicine (RITM)
Locations (1):
- Research Institute for Tropical Medicine (RITM), Alabang, Muntinlupa City, Philippines

REFERENCES:
- [Result] Bhutta ZA, Capeding MR, Bavdekar A, Marchetti E, Ariff S, Soofi SB, Anemona A, Habib MA, Alberto E, Juvekar S, Khan RM, Marhaba R, Ali N, Malubay N, Kawade A, Saul A, Martin LB, Podda A. Immunogenicity and safety of the Vi-CRM197 conjugate vaccine against typhoid fever in adults, children, and infants in south and southeast Asia: results from two randomised, observer-blind, age de-escalation, phase 2 trials. Lancet Infect Dis. 2014 Feb;14(2):119-29. doi: 10.1016/S1473-3099(13)70241-X. Epub 2013 Nov 28. PMID 24290843

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Started | 20 | 20 | 20 | 20 | 20 | 20
Completed | 20 | 19 | 20 | 19 | 20 | 20
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20 | 120
Age, Customized [Number; unit: participants]
  6 weeks to 8 weeks (infants) | 0 | 0 | 0 | 0 | 20 | 20 | 40
  9 months to 12 months (older infants) | 0 | 0 | 20 | 20 | 0 | 0 | 40
  24 months 59 months (children) | 20 | 20 | 0 | 0 | 0 | 0 | 40
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 12 | 14 | 11 | 10 | 69
  Male | 8 | 10 | 8 | 6 | 9 | 10 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 20 | 20 | 20 | 20 | 20 | 20 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Philippines | 20 | 20 | 20 | 20 | 20 | 20 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi Enzyme-linked Immunosorbent Assay (ELISA) Titer
Time Frame: At 28 days after last vaccination as compared to baseline
Population: Intention-to-treat analysis set, which included all participants who received the vaccination, those in whom at least one post-vaccination blood sample was collected, and those for whom at least one ELISA result was available.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 20 | 19 | 20 | 19 | 20 | 20
percentage of subjects | 100 [83 to 100] | 100 [82 to 100] | 100 [83 to 100] | 11 [1 to 33] | 100 [83 to 100] | 10 [1 to 32]

2. Primary Outcome: Percentage of Subjects With at Least 4-fold Increase in Anti-Vi ELISA Titer
Time Frame: At 6 months after last vaccination as compared to baseline
Population: Intention-to-treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 20 | 19 | 20 | 19 | 20 | 20
percentage of subjects | 90 [68 to 99] | 95 [74 to 100] | 70 [46 to 88] | 11 [1 to 33] | 70 [46 to 88] | 5 [0 to 25]

3. Primary Outcome: Anti-Vi ELISA Geometric Mean Concentration (GMC)
Time Frame: At 28 days after last vaccination
Population: Intention-to-treat analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 20 | 19 | 20 | 19 | 20 | 20
ELISA Units/mL | 255 [174 to 375] | 107 [72 to 159] | 129 [83 to 200] | 3.79 [2.41 to 5.97] | 103 [67 to 159] | 5.05 [3.27 to 7.79]

4. Primary Outcome: Anti-Vi ELISA GMC
Time Frame: At 6 months after last vaccination
Population: Intention-to-treat analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units/mL
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 20 | 19 | 20 | 19 | 20 | 20
ELISA Units/mL | 51 [34 to 76] | 45 [30 to 68] | 21 [14 to 31] | 3.69 [2.41 to 5.65] | 21 [16 to 28] | 2.64 [1.98 to 3.52]

5. Secondary Outcome: Number of Participants With Any Solicited Local and Systemic Reaction, After Any Vaccination
Description: Solicited local reactions were: erythema, induration, pain/tenderness. Solicited systemic reactions were; lethargy, irritability, vomiting, diarrhoea, loss of appetite (and persistent crying in the older infants and infants age group)
Time Frame: During the 7-day follow-up period after vaccination
Population: Analysis was done on as treated safety population
Measure: Number; unit: participants
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 20
participants | 11 | 10 | 12 | 17 | 20 | 19

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events (AEs) were collected during 7-day follow period after each vaccination. Serious AEs were collected throughout the study period. Unsolicited AEs were collected collected during 28-day follow period after each vaccination.
Arm/Group | Vi-CRM, Children | Vi-PS, Children | Vi-CRM, Older Infants | PNC13, Older Infants | Vi-CRM, Infants | PNC13, Infants
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20 | 0/20 | 0/20 | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 14/20 | 14/20 | 17/20 | 20/20 | 20/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vi-CRM, Children (N=20) | Vi-PS, Children (N=20) | Vi-CRM, Older Infants (N=20) | PNC13, Older Infants (N=20) | Vi-CRM, Infants (N=20) | PNC13, Infants (N=20)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vi-CRM, Children (N=20) | Vi-PS, Children (N=20) | Vi-CRM, Older Infants (N=20) | PNC13, Older Infants (N=20) | Vi-CRM, Infants (N=20) | PNC13, Infants (N=20)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 6 | 6 | 4 | 6
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5 | 4 | 5 | 5
Crying (General disorders) | 0 | 0 | 1 | 4 | 13 | 12 — systemic assessment for older infants and infants
Induration (General disorders) | 0 | 0 | 0 | 0 | 7 | 3
Injection site erythema (General disorders) | 1 | 2 | 5 | 11 | 12 | 8
Injection site induration (General disorders) | 2 | 2 | 1 | 5 | 14 | 15
Injection site pain (General disorders) | 6 | 7 | 3 | 10 | 20 | 18
Irritability (General disorders) | 1 | 2 | 2 | 6 | 12 | 14
Pyrexia (General disorders) | 3 | 4 | 7 | 10 | 7 | 8
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 4 | 6 | 3
Impetigo (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Mumps (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 6 | 3 | 4 | 4
Respiratory tract infections (Infections and infestations) | 0 | 1 | 1 | 2 | 3 | 3
Rhinitis (Infections and infestations) | 1 | 0 | 4 | 3 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 7 | 5 | 6 | 9 | 10
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2 | 4 | 8 | 10
Eating disorders (Psychiatric disorders) | 0 | 2 | 2 | 8 | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event that no publication of the Study results has been made by NVGH within twelve (12) months of Study database lock and no proposed publication is under discussion by the publication committee, Principal Investigator may publish its own Study results.